CLINICAL TRIAL: NCT01050296
Title: Molecular Analysis Of Solid Tumors
Acronym: MAST
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Alex's Lemonade Stand Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: MAST; DOD-W81XWH-14-1-0103(CA130396) (Other Grant/Funding Number: DOD-Department of the Army)
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Solid Tumors
Keywords: Neuroblastoma; Retinoblastoma; Osteosarcoma; Rhabdomyosarcoma; Ewing sarcoma; Non-rhabdomyosarcoma soft tissue sarcoma; Adrenocortical tumors; Liver malignancies
MeSH Terms: conditions — Neuroblastoma; Retinoblastoma; Osteosarcoma; Rhabdomyosarcoma; Sarcoma, Ewing; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue - Tumor tissue will be obtained from patients with a diagnosis of neuroblastoma, retinoblastoma, osteosarcoma, Ewing sarcoma or soft tissue sarcoma at some or all of the following time points: initial biopsy, primary tumor resection, time of disease recurrence. Whole blood - 5 ml of whole blood will be collected from each patient and be used as a matched control. Bone marrow aspiration - 5ml of bone marrow will be taken at the time a patient is having a bone marrow aspirate performed and processed to remove only tumor cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will prospectively characterize the molecular, cellular and genetic properties of primary and metastatic neuroblastoma, osteosarcoma, retinoblastoma, Ewing sarcoma family of tumors, soft tissue sarcomas, adrenocortical tumors and liver malignancies. These cell isolates will be used for gene expression array analysis, genomic analysis by [SNP] single nucleotide polymorphism chip, array [CGH] comparative genomic hybridization and next generation sequencing, and [TEM] transmission electron microscopy analysis. Additionally cell lines and orthotopic xenografts will be created from the obtained tumor specimens.

The specificity of TCRs will be examined by comparing paired TCR from peripheral blood and tumor infiltrating CD4+ and CD8+ T cells. Epigenetic studies will be performed looking at the methylation profile of these cells and to investigate the anti-tumor T cell response both pre- and post-PD1 inhibition.

DETAILED DESCRIPTION:
Each year approximately 2,200 children in the United States are diagnosed with neuroblastoma, osteosarcoma, Ewing sarcoma family of tumors (ESFT), retinoblastoma, soft tissue sarcomas, adrenocortical tumors and liver malignancies. These aggressive pediatric solid tumors are developmental tumors that initiate during periods of tissue growth and morphogenesis in the neural crest, bone and soft tissues. The overall survival rate of these tumors in the advanced stage is less than 30%. Despite intensive efforts over the past three decades using multiple therapeutic modalities including chemotherapy, surgery, radiation, autologous bone marrow transplant and biological agents there has been modest improvement in the long-term survival of these advanced stage pediatric solid tumors. A better understanding of the molecular, cellular and genetic changes that occur in the developing tissues as tumors form could improve the treatment of these devastating cancers. In particular, chemotherapeutic agents may be more effectively targeted to key regulatory enzymes or proteins if the study had a better understanding of the pathways that are disrupted as cells progress from preneoplastic lesions to metastatic disease. The specific aim of this proposal is to identify the changes in gene expression that occur in neuroblastoma, retinoblastoma, osteosarcoma, Ewing sarcoma family of tumors [ESFT] and soft tissue sarcoma cells and to correlate these changes with genetic and cellular changes in the tumor cells. [RNA] ribonucleic acid and genomic [DNA] deoxyribonucleic acid will be isolated from neuroblastoma, retinoblastoma, osteosarcoma, ESFT [Ewing sarcoma family of tumors] and soft tissue sarcomas (both primary and metastatic lesions) following surgery or bone marrow aspiration of previously untreated patients. Additional testing will be conducted on tumor samples at any point during or following therapy in which a surgical specimen is obtained. When there is sufficient tumor sample remaining after pathological analysis and banking, fresh primary tumor cells will be used to prepare orthotopic xenografts and to establish models of each disease that recapitulate the advanced forms of neuroblastoma, osteosarcoma, Ewing sarcoma family of tumors [ESFT], retinoblastoma and soft tissue sarcomas. For a small group of these excess samples, this study will perform fixation for electron microscopy and process the samples for [TEM] transmission electron microscopy analysis. These studies will complement our active research program characterizing the molecular, cellular and genetic features of genetically engineered mouse models of each of these diseases. Biological samples from the cohort of patients treated at St. Jude Children's Research Hospital will be complemented with samples collected and processed by collaborating institutions around the world. Samples collected from international collaborators will be used for analysis of [DNA] deoxyribonucleic acid and [RNA] ribonucleic acid to complement the St. Jude Children's Research Hospital cohort. Through this collaboration the study anticipates that they will be able to obtain enough fresh tumor samples to improve their understanding of multistage tumorigenesis in pediatric solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Must have a suspected or known diagnosis of neuroblastoma, osteosarcoma, Ewing sarcoma family of tumor or soft tissue sarcoma based on the initial diagnostic workup and evidence of gross disease amenable to excision. Specimens may be collected at some or all of the following time points: initial biopsy, bone marrow aspiration procedures, tumor resection, and at time of possible relapse.
* Patients with a diagnosis of retinoblastoma based on initial diagnostic workup and who require enucleation may be enrolled if there is no active therapeutic or biologic protocol for retinoblastoma.
* The patient or his/her legal guardian, as appropriate, must provide written informed consent within 30 days of the removal of the first collection of tissue/bone marrow/blood sample for this protocol.
* The patient is being seen at St. Jude Children's Research Hospital or at a collaborating institution.
* Patients must be less than or equal to 25 years old at the time of enrollment.

Exclusion Criteria:

* Patient is known to be Hepatitis B, Hepatitis C and/or HIV positive.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients identified at St. Jude Children's Research Hospital and collaborating institutions with a suspected or known diagnosis of neuroblastoma, osteosarcoma, retinoblastoma, Ewing sarcoma or soft tissue sarcoma based initial diagnostic workup and evidence of gross disease amenable to excision.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-02-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Perform analysis of gene expression profiles. [RNA] ribonucleic acid will be isolated from fresh frozen tumor specimens and hybridized to Affymetrix gene expression arrays. | 5 years

SECONDARY OUTCOMES:
Perform analysis of large chromosomal alterations such as amplifications and deletions. [DNA] deoxyribonucleic acid isolated from the tumor and blood samples will be hybridized to array [CGH] comparative genomic hybridization chips. | 5 years
Perform analysis of focal alterations in the genome including amplification, deletion and loss of heterozygosity (LOH). DNA isolated from the tumor and blood samples will be hybridized to [SNP] single nucleotide polymorphism chips. | 5 years
Perform analysis of point mutations. DNA isolated from the tumor and blood samples will be sequenced using next-generation sequencing technology to determine the sequence of the entire genome. | 5 years
Perform analysis of cell morphology. Tissue samples will be fixed in a buffer suitable for transmission electron microscopy and processed for [TEM] transmission electron microscopy analysis. | 5 years
Compare micro RNAs in tumors. Micro RNAs will be isolated from the total [RNA] ribonucleic acid left over from the gene expression analysis described above. These samples will be used for micro [RNA] chip analysis or deep sequencing. | 5 years
Compare epigenetic modifications of [DNA] deoxyribonucleic acid. Genomic DNA will be isolated and DNA methylation will be analyzed across the genome to determine if this epigenetic process is altered in the tumor samples. | 5 years
Compare epigenetic modifications of chromatin. Cells will be rapidly fixed and chromatin will be prepared in order to directly probe protein-DNA complexes by [ChIP-seq]chromatin immunoprecipitation or [ChIP-chip analysis] chromatin immunoprecipitation | 5 years
Perform protein analysis. Tumor cells will be rapidly frozen for subsequent isolation of total protein or specific fraction of cellular proteins (i.e. nuclear, cytoplasmic, membrane proteins). | 5 years
Perform immunohistochemical and FISH analysis of neuroblastoma, osteosarcoma, retinoblastoma, ESFT and soft tissue sarcomas. Tissue microarrays will be prepared from samples collected in this study. | 5 years
Cell isolates obtained from primary and metastatic tumor specimens will be used to establish cell lines and orthotopic xenografts in immunocompromised mice. | 5 years
Perform analysis of cell growth, metastasis and sensitivity to chemotherapy. | 5 years
Evaluate the extent of immune cell infiltration and their functional status in pediatric solid tumors utilizing flow cytometric analysis of fresh tumor samples. | 5 years
Evaluate tumor-associated macrophages (TAMSs) post-therapy to locate gene expression patterns, markers and functional correlates of the tissue repair properties of macrophages in the post-therapy microenvironment. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sara M. Federico, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols